CLINICAL TRIAL: NCT01840371
Title: Randomized Controlled Study for Analyzing Clinical Benefit of Pain Focused Sedation With Combination of Fentanyl and Propofol During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 4-2013-0012
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; Sedation; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol based group (Experimental)
  Interventions: Drug: Conventional sedation
- Fentanyl based group (Active Comparator)
  Interventions: Drug: Experimental sedation

INTERVENTIONS:
Drug: Conventional sedation — Propofol Meperidine : 25 mg IV just before procedure
  * IV bolus of 1 mg/kg for sedation induction,
  * Infusion of 60 mcg/min/kg for maintenance of sedation
  * Additional bolus dose of 10mg as needed for adequate sedation
  Arms: Propofol based group
Drug: Experimental sedation — Fentanyl
  * IV bolus of 1 µg/kg for sedation induction
  * Additional bolus dose of 0.5 µg/kg as needed for adequate pain control Propofol
  * IV bolus of 0.4 mg/kg for sedation induction
  * Infusion of 30 µg/min/kg for maintenance of sedation
  * Additional bolus dose of 10mg as needed for adequate depth of sedation
  Arms: Fentanyl based group

SUMMARY:
The investigators study is the randomized controlled study for analyzing clinical benefit of pain focused sedation with combination of fentanyl and propofol during Endoscopic retrograde cholangiopancreatography (ERCP). The investigators will assess recovery time and adverse effect during ERCP as the primary end point between two group. The investigators will also access satisfaction score for endoscopist and patients as the secondary end point.

ELIGIBILITY:
Inclusion Criteria:

* The patients who scheduled for ERCP

Exclusion Criteria:

* The patients with ASA physical classification V
* The patients with history of sulfite, egg or soy bean allergy
* The patients during pregnancy or latency period
* The patients who informed consent could not be obtained
* The patients who were under 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Recovery time | time from scope withdrawal to full recovery at averange 24 hours
  Recovery time (time from scope withdrawal to full recovery)

SECONDARY OUTCOMES:
Adverse event during and after procedure | measurements of recovery time during ERCP procedure & after ERCP procedure at average 24 hours
  Adverse event during and after procedure i. Desaturation rate ii. Apnea

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, Seoul, South Korea

REFERENCES:
- [Result] Lee TH, Lee CK, Park SH, Lee SH, Chung IK, Choi HJ, Cha SW, Moon JH, Cho YD, Hwangbo Y, Kim SJ. Balanced propofol sedation versus propofol monosedation in therapeutic pancreaticobiliary endoscopic procedures. Dig Dis Sci. 2012 Aug;57(8):2113-21. doi: 10.1007/s10620-012-2234-0. Epub 2012 May 22. PMID 22615018
- [Result] Angsuwatcharakon P, Rerknimitr R, Ridtitid W, Kongkam P, Poonyathawon S, Ponauthai Y, Sumdin S, Kullavanijaya P. Cocktail sedation containing propofol versus conventional sedation for ERCP: a prospective, randomized controlled study. BMC Anesthesiol. 2012 Aug 9;12:20. doi: 10.1186/1471-2253-12-20. PMID 22873637